CLINICAL TRIAL: NCT03038750
Title: Molecular Investigation of Genetic Factors in CArDiovascular Diseases Using an BIOresource of Healthy Volunteers
Acronym: CADBIO
Status: Terminated | Type: Observational
Why Stopped: The delay due to suspending the study due to covid, subsequent problems in synthesis, supply and yield of BQ123, prevented completion of the study as planned.
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: University of Cambridge (Other)
Responsible Party: Principal Investigator, Dirk Paul, Principal Investigator, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: CADBIO
Record Dates: First submitted 2017-01-25; First posted 2017-02-01 (Estimated); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Cardiovascular Diseases
Keywords: Healthy Volunteers; Genetic Risk Markers for Cardiovascular Disease; Non-Alcoholic Fatty Liver Disease; Coronary Disease; Hypertension; Venous Thromboses; Venous Thromboembolism; Coronary Heart Disease; Coronary Artery Disease
MeSH Terms: conditions — Cardiovascular Diseases; Non-alcoholic Fatty Liver Disease; Coronary Disease; Hypertension; Venous Thrombosis; Venous Thromboembolism; Coronary Artery Disease | interventions — Eligibility Determination; Health Records, Personal; Demography; Weights and Measures; Blood Pressure; Heart Rate; Receptor, Endothelin A; adiponutrin; Endothelial Protein C Receptor; Functional Status; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- EDNRA Sub-study: Study population will be split into two groups defined by the allele of EDNRA the participant possesses:
  Participants Homozygous for the A-allele of EDNRA, are assigned to the 'case' group.
  Participants that are Homozygous for the G-allele will be assigned to the 'control' group.
  20 participants will be recruited to each group, 40 in total.
  Interventions: Other: Eligibility and lifestyle restrictions check.; Other: Medical history, demographic and lifestyle factors; Other: Anthropometric measurements: height, weight, and body fat; Other: Blood pressure and heart rate; Other: Forearm blood flow: Visit 1 (EDNRA); Other: Forearm blood flow: Visit 2 (EDNRA)
- PNPLA3 Sub-study: Study population will be split into two groups defined by the allele of PNPLA3 the participant possesses:
  Participants Homozygous for the G-allele of PNPLA3, are assigned to the 'case' group.
  Participants that are Homozygous for the C-allele of PNPLA3 will be assigned to the 'control' group.
  60 participants will be recruited to each group, 120 in total.
  Interventions: Other: Eligibility and lifestyle restrictions check.; Other: Medical history, demographic and lifestyle factors; Other: Anthropometric measurements: height, weight, and body fat; Other: Blood pressure and heart rate; Other: Blood biochemistry (PNPLA3); Other: Baseline Venepuncture (PNPLA3, Visit 1); Other: Deuterium water - Loading dose 1 (PNPLA3, Visit 1); Other: Deuterium water - Loading dose 2 (PNPLA3, Visit 1); Other: Energy-balanced dinner (PNPLA3, Visit 1); Other: Fasting venepuncture (PNPLA3, Visit 2); Other: Deuterium water - Maintenance dose (PNPLA3, Visit 2); Other: Consumption of high carbohydrate meal (PNPLA3, Visit 2); Other: Postprandial Venepuncture (PNPLA3, Visit 2)
- PROCR Sub-study: Study population will be split into two groups defined by the allele of PROCR the participant possesses:
  Participants Homozygous for the G-allele of PROCR, are assigned to the 'case' group.
  Participants that are Homozygous for the A-allele of PROCR will be assigned to the 'control' group.
  30 participants will be recruited to each group, 60 in total.
  Interventions: Other: Eligibility and lifestyle restrictions check.; Other: Medical history, demographic and lifestyle factors; Other: Anthropometric measurements: height, weight, and body fat; Other: Blood pressure and heart rate; Other: Blood EPCR function (PROCR); Other: Blood platelet coagulation and function (PROCR); Other: Blood endothelial permeability (PROCR); Other: Blood leukocyte-endothelium adhesion (PROCR); Other: Venepuncture (PROCR)

INTERVENTIONS:
Other: Eligibility and lifestyle restrictions check. — Eligibility will be assessed at each study visit and participants will be informed in advance of their visit.
Other: Medical history, demographic and lifestyle factors — Medical History, participants demographics and lifestyle factors will be assessed by the participant completion of the medical history and ethnicity questionnaires.
Other: Anthropometric measurements: height, weight, and body fat — Height measured by stadiometer. Weight and body fat measured by Tanita scale bioelectrical impedance analysis.
Other: Blood pressure and heart rate — Parameters will be measured using a validated, automated device while seated and again after 3-5 min standing. All measurements will be done in triplicate.
Other: Forearm blood flow: Visit 1 (EDNRA) — Intra-arterial infusion of Phenylephrine at doses of 0.75, 2.5, and 7.5 μg/min for 6 min each (18 min in total). FBF measured in the last 3 minutes. There will be a 30 minute washout with saline followed by Endothelin-1 infusion of at a dose of 5 pmol/min for 90 min.
  Groups: EDNRA Sub-study
Other: Forearm blood flow: Visit 2 (EDNRA) — Intra-arterial infusion of Sodium nitroprusside infusion at doses of 1, 3, and 10 μg/min for 6 min each (18 min in total). FBF measured in the last 3 minutes. There will be a 20 minute washout with saline followed by infusion of BQ-123 at a dose of 10 nmol/min for 90 min.
  Groups: EDNRA Sub-study
Other: Blood biochemistry (PNPLA3) — 25ml blood will be taken from the participant in a glucose fasting state. Following a high carbohydrate meal, a second 25ml blood sample will be taken. Clinical Biochemistry tests and detailed lipid analysis will be performed.
  Groups: PNPLA3 Sub-study
Other: Blood EPCR function (PROCR) — Blood sample taken will be analysed via ELISA and FACS.
  Groups: PROCR Sub-study
Other: Blood platelet coagulation and function (PROCR) — Blood sample taken will be analysed using a Platelet coagulation and function assay.
  Groups: PROCR Sub-study
Other: Blood endothelial permeability (PROCR) — Blood sample will be analysed in vitro using a permeability assay kit.
  Groups: PROCR Sub-study
Other: Blood leukocyte-endothelium adhesion (PROCR) — Blood sample will be analysed in vitro using a leukocyte-endothelium adhesion assay.
  Groups: PROCR Sub-study
Other: Baseline Venepuncture (PNPLA3, Visit 1) — Up to 25ml Blood will be taken.
  Groups: PNPLA3 Sub-study
Other: Deuterium water - Loading dose 1 (PNPLA3, Visit 1) — Loading dose of 3 g/kg body water.
  Groups: PNPLA3 Sub-study
Other: Deuterium water - Loading dose 2 (PNPLA3, Visit 1) — Loading dose of 3 g/kg body water.
  Groups: PNPLA3 Sub-study
Other: Energy-balanced dinner (PNPLA3, Visit 1) — Provided following baseline bloods and loading dose 1.
  Groups: PNPLA3 Sub-study
Other: Fasting venepuncture (PNPLA3, Visit 2) — Up to 25ml Blood will be taken.
  Groups: PNPLA3 Sub-study
Other: Deuterium water - Maintenance dose (PNPLA3, Visit 2) — every hour, maintenance dose 0.04 g/kg body water
  Groups: PNPLA3 Sub-study
Other: Consumption of high carbohydrate meal (PNPLA3, Visit 2) — Provided following fasting blood sample.
  Groups: PNPLA3 Sub-study
Other: Postprandial Venepuncture (PNPLA3, Visit 2) — Up to 25ml Blood will be taken.
  Groups: PNPLA3 Sub-study
Other: Venepuncture (PROCR) — Up to 50ml Blood will be taken.
  Groups: PROCR Sub-study

SUMMARY:
The risk of cardiovascular disease is determined by the complex interplay between an individual's genetic make-up, lifestyle, and the environment. We are investigating three potential genetic risk factors in this observational, cross-sectional, epidemiology pilot study to investigate if and how functional variants identified in large-scale genome wide association studies can explain a predisposition to cardiovascular disease. By determining the molecular mechanisms that are regulated at the EDNRA, PNPLA3 and PROCR CVD risk loci, we hope to translate findings from this study into the clinical setting for better diagnosis, prevention and treatment for patients suffering with cardiovascular disease. Volunteers will enter into one of the study's three arms based on their genotype: EDNRA locus (Arm 1), PNPLA3 locus (Arm 2), or PROCR locus (Arm 3).

Members of the Cambridge Bioresource who match for the target alleles will be invited to participate and will enter into one of the three study arms. All study assessment visits will take place at Addenbrooke's Hospital in collaboration with the University of Cambridge.

Volunteers will participate in the study for a maximum of 12 months and depending on study arm they are assigned to, they will complete procedures including a medical, demographic and lifestyle factors questionnaire; height, weight and body fat assessments; in addition to blood pressure/heart rate measurements. Minimally invasive procedures including forearm blood flow and venepuncture will be performed to assess the primary objectives of the study.

The hypothesis for arm 1 is that the genetic variant we are investigating at the EDNRA gene locus alters the function of the endothelin receptor A leading to an increased risk of coronary artery disease and large artery stroke.

For study arm 2, we hypothesize that the genetic variant we are investigating in PNPLA3 will increase the risk of Non-alcoholic fatty liver disease but reduce the risk of Coronary Heart Disease.

For study arm 3, we hypothesize that the genetic variant we are investigating in the PROCR locus triggers molecular events that potentially increase the risk of Venous Thrombosis/Venous Thromboembolism nut reducing blood pressure. Furthermore we aim to investigate the anti-inflammatory effects to see if there is an effect on explaining reduced risk of CHD.

This study is funded from the BHF Cambridge Center of Excellence and the Wellcome Trust Institutional Strategic Support Fund.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers are homozygous for:

  * Arm 1: The A-allele of rs6841581, they are assigned to the 'case' group. If they are homozygous for the G-allele, they are assigned to the 'control' group
  * Arm 2: The G-allele of rs738409, they are assigned to the 'case' group. If they are homozygous for the C-allele, they are assigned to the 'control' group
  * Arm 3: The G-allele of rs867186, they are assigned to the 'case' group. If they are homozygous for the A-allele, they are assigned to the 'control' group
* Volunteers are aged between 18-50 years old
* Volunteers have a BMI:

  * Arm 1: Between18.5-29.9
  * Arm 2: Between 25.0-39.9
  * Arm 3: Between 18.5-29.9
* Volunteers are willing not to consume products containing alcohol or caffeine 12 hours prior to procedures. Additionally, volunteers must agree to fast before procedures for:

  * Arm 1: At least 4 hours
  * Arm 2: At least 8 hours (for visit 2 only)
  * Arm 3: At least 4 hours
* Have given written informed consent to participate

Exclusion Criteria:

* Volunteers with chronic diseases, including cardiovascular diseases, liver diseases, type 1 and type 2 diabetes autoimmune diseases and cancer
* Biological first-degree relatives (parents, brothers, sisters or children) who are or have suffered from one of the conditions described above
* Current smokers. Ex-smokers are suitable if they stopped smoking >10 years ago
* Volunteers with a diagnosis of hypertension, or history of consistently high blood pressure readings, >140/90 mmHg
* Volunteers with a diagnosis of hypercholesterolemia, or history of consistently high cholesterol levels, e.g. total cholesterol level >6 mmol/l
* Volunteers have ≥3 alcoholic drinks per day

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will only recruit healthy volunteers who have previously consented to being contacted for future studies by the NIHR Cambridge BioResource which is a panel of around 20,000 volunteers, both with and without health conditions, who are willing to be approached to participate in research studies investigating the links between genes, the environment, health and disease. Volunteers who join the Cambridge BioResource have donated their DNA via a blood or saliva sample which is used together with other information, such as gender and ethnicity, to match them to specific research studies. Participants for this study are therefore identified by having the appropriate genetic sequence in one of the three genetic loci we are investigating (EDNRA, PNPLA3 or PROCR).
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Forearm Blood Flow (Arterial contractility) | 2 years
  Arm 1 specific measurement to be measured using venous occlusion plethysmography. Outcome measure will compare results between case vs control groups.
Blood Biochemistry (Lipoprotein composition/dynamics) | 2 years
  Arm 2 specific measurement collectively comparing the lipid dynamic results between case vs control groups.
EPCR levels/shedding | 2 years
  Arm 3 specific measurement comparing results between case vs control groups.
Platelet aggregation/function | 2 years
  Arm 3 specific measurement to be measured by platelet coagulation function assay comparing results between case vs control groups.
Endothelial permeability | 2 years
  Arm 3 specific measurement to be measured by an endothelial permeability assay comparing results between case vs control groups.
Leukocyte-endothelium adhesion | 2 years
  Arm 3 specific measurement to be measured by a leukocyte-endothelium adhesion assay comparing results between case vs control groups.

SECONDARY OUTCOMES:
Blood pressure | 2 years
  All study arms comparing results between case vs control groups.
Heart rate | 2 years
  All study arms comparing results between case vs control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Paul, PhD, Principal Investigator — University of Cambridge
Locations (1):
- Department of Public Health and Primary Care, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Participant identifiable information is securely held, with restricted access, by the NIHR BioResource. Members of the research team carrying out the procedures will not be able to request the link to decode this information. Only the minimum required participant identifiable information (name and contact details) will be provided to the research team for the purpose of arranging study visits and completing the informed consent process. All research personnel will be sufficiently blinded of the genotype status of the healthy volunteers. All delegated research personnel that is responsible to conduct the data/statistical analysis will only analyse data that is anonymised of any patient identifiable data.